CLINICAL TRIAL: NCT05416437
Title: Breathlessness Relieved by Employing Medical Air to be Titrated by Hospitalized Patients to Improve Inpatient Experience
Acronym: BREATHE-easy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Sonal Pannu, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021H0334
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Masking Description: The is an open label study. There is no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device arm (Active Comparator): The patients in the device arm will get the Pneumocool device to channel medical air to their face to alleviate dyspnea
  Interventions: Device: PneumoCool
- Standard of Care arm (Placebo Comparator): The patients in the standard of care arm can get a fan or any other supportive care that is currently available in the hospital for alleviating dyspnea
  Interventions: Other: Current supportive measures that are used in the hospital for standard of care

INTERVENTIONS:
Device: PneumoCool — Device to channel medical air to the patient to alleviate dyspnea
  Arms: Device arm
Other: Current supportive measures that are used in the hospital for standard of care — a room fan, or any other currently used supportive measures can be used for patients in the control arm
  Arms: Standard of Care arm

SUMMARY:
The BREATHE-easy is a randomized control trial assessing the efficacy of the novel PneumoCool device to alleviate subjective shortness of breath. The PneumoCool device is a disposable, bladeless, highly portable device that uses medical-grade air that confers many advantages in a hospital setting.

DETAILED DESCRIPTION:
This will be randomized control trial (RCT) for patients admitted to the Ohio State University Wexner Medical Center, ROSS and James Cancer Hospital. Patients will be screened to assess eligibility. The study team will use a 2-group (intervention vs. control) RCT design. On meeting inclusion criteria, completed informed consent will be obtained. After informed consent, subjects will be randomized to receive either the PneumoCool device or usual therapy. PneumoCool setup will be done by the study team. This study will be unblinded, since blinding is not feasible in this device study. Conventional therapy will include the patients usual care and any palliation for patients' symptoms ordered by the primary team, including bedside fan if the patient requests. Patients will be queried for their symptoms at the time of enrollment, at time 0 (start of first arm of trial) and 8 hours for the primary outcome. Patient will be followed throughout their hospital stay until discharge. Data will be collected from the electronic medical record. Patient and Provider satisfaction will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Dyspnea (Borg Scale > 3)
* Admitted to University hospital, ROSS or James Cancer Hospital with expected length of stay > 24 hours
* Age 18 years or more

Exclusion Criteria:

* Delirium (assessed by CAMICU) or dementia or brain injury precluding ability to consent and or respond to outcome scales
* Prisoner status
* Continuous mechanical ventilation
* Patients with motor disability with inability to maneuver the device

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Borg Dyspnea scale ( (0 indicating no effort of breathing, 10 indicating maximal effort of breathing) | At 8 hours after enrollment
  Mean changes in the Borg Dyspnea scale (0 indicating no effort of breathing, 10 indicating maximal effort of breathing)

SECONDARY OUTCOMES:
Visual analog scale (0 indicating no trouble breathing, 10 indicating severe shortness of breath) | At 8 hours after enrollment
  Mean Change visual analog scale
Supplemental oxygen | At 48 hours after study enrollment
  change of supplemental oxygen
External cooling devices | From enrollment to hospital discharge or 30 days whichever happens earlier
  Duration of external cooling devices (hours)
Bronchodilator dosage | At 48 hours after study enrollment
  Mean changes in Bronchodilator doses
Benzodiazepine dosage | At 48 hours after study enrollment
  Mean changes in Benzodiazepine doses
Opoid dosage | At 48 hours after study enrollment
  Mean changes in Opoid doses
Bedside provider calls for dyspnea | At 48 hours after study enrollment
  Mean changes in bedside provider calls for dyspnea
Need for Noninvasive positive pressure ventilation [NIPPV] or Invasive mechanical ventilation) | Upto hospital discharge or death which every happens earlier upto 60 day after enrollment
  Note the need for Noninvasive positive pressure ventilation [NPIIV] or Invasive mechanical ventilation
Hospital length of stay | Upto hospital discharge or death which every happens earlier upto 60 day after enrollment
  Note duration of hospitalization
ICU length of stay | Upto transfer from ICU or death which every happens earlier upto 60 day after enrollment
  Note duration of ICU stay for those patients in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Sonal R Pannu, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No